CLINICAL TRIAL: NCT05292924
Title: Immediate vs Early Skin-to-skin Contact in Cesarean Births and Its Effect on Breastfeeding
Brief Title: Early Versus Inmediately Skin to Skin Contact in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asociación Mexicana de Salud Primal (Other)
Responsible Party: Principal Investigator, Jose Octavio Zavala Soto, Doctorate of social sciences, Asociación Mexicana de Salud Primal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Skin-to-Skin-cesarean
Record Dates: First submitted 2022-03-15; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Breastfeeding, Exclusive; Mother-Child Relations; Kangaroo-mother Care
Keywords: Birth; Cesarean Section; Skin-to-skin contact; Mother-Child Relations; Breastfeeding; kangaroo-mother care
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: 6000 births per year were considered, of which 30% correspond to births by cesarean section. For a non-random and voluntary sampling with a homogeneous population and a sampling error of 5%, at a confidence level of 95%, the sample size is 278. Of this number of participants, 50% will be assigned to the experimental group (birth by cesarean section and EFS within the first 30 minutes of birth) and 50% to the control group (caesarean birth and EFS one hour after birth) by simple randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early SSC (Experimental): Cesarean delivery and SSC within the first 30 minutes of birth
  Interventions: Procedure: Early SCC
- Control (No Intervention): Cesarean delivery and SSC one hour after birth

INTERVENTIONS:
Procedure: Early SCC — Direct, immediate and uninterrupted contact of the infant with its mother's skin first 30 minutes delivery
  Arms: Early SSC

SUMMARY:
Breastfeeding plays a fundamental role in the health of girls and boys by providing adequate nutrition, promoting development and mainly preventing diseases. Different maternal factors such as education or obesity and perinatal factors such as the route of birth or skin-to-skin contact, among many others, can influence its onset, proper establishment and duration. Caesarean section and instrumental delivery are directly related to a delay in the early initiation of breastfeeding in newborns. In Mexico, the rate of caesarean sections is well above that recommended by the World Health Organization, in addition to being a country with very low rates of exclusive breastfeeding at 6 months of age of the newborn without having achieved the proposed objectives to improve it in recent years.

Newborns who experience skin-to-skin contact with their mother develop behaviors such as crawling to the breast and more effective suckling with greater lactogenesis by the mother. The World Health Organization (WHO) defines skin-to-skin contact (SSC) as "direct, immediate and uninterrupted contact of the infant with the mother's skin" and promotes it because it is important for establishment of breastfeeding, neonatal and child survival and development. It has been seen that the ideal time to start this CPP is within the first 30 minutes of life of the newborn in any birth route, so it has been recommended that it be started in the recovery room or even in the operating room during birth by caesarean section in order to make a mark in the programming of the future physiology and behavior of the dyad.

The foregoing leads us to ask ourselves the following research questions: Can we in our public hospitals in Mexico carry out the CPP procedure between mother and baby during cesarean births? And if so, will there be a difference in breastfeeding by Mexican women, performing skin-to-skin contact immediately even in the operating room between mother and baby in cesarean births versus if it is carried out after the surgical procedure?

DETAILED DESCRIPTION:
Breastfeeding plays a fundamental role in the health of girls and boys by providing adequate nutrition, promoting development and mainly preventing diseases. Different maternal factors such as education or obesity and perinatal factors such as the route of birth or skin-to-skin contact, among many others, can influence its onset, proper establishment and duration. Caesarean section and instrumental delivery are directly related to a delay in the early initiation of breastfeeding in newborns. The cause of this effect has been related to the limitation in maternal movement, the pain of the wound or the difficulty in maternal positioning. It has also been seen that newborns by caesarean section or instrumental delivery may have more problems with attachment and inadequate suction. In Mexico, the rate of caesarean sections is well above that recommended by the World Health Organization, in addition to being a country with very low rates of exclusive breastfeeding at 6 months of age of the newborn without having achieved the proposed objectives to improve it in recent years.

Cesarean section traditionally implies a separation between the mother and her newborn, which is contrary to the recommendations to promote better breastfeeding and establishment of the bond between the mother and her baby. There is evidence that demonstrates the relationship between skin-to-skin contact and higher rates of exclusive breastfeeding. This contact between the naked baby on the naked torso of her mother as soon as possible after birth is also recommended in cesarean births as soon as possible for the mother to perform it.

Newborns who experience skin-to-skin contact with their mother develop behaviors such as crawling to the breast and more effective suckling, in addition to having the opportunity to manifest the necessary demands for attention that trigger neuropsychobiological pathways that activate maternal behaviors and a immediate response to the needs of the infant with greater lactogenesis by the mother. The World Health Organization (WHO) defines skin-to-skin contact (SSC) as "direct, immediate and uninterrupted contact of the infant with the mother's skin" and promotes it because it is important for establishment of breastfeeding, neonatal and child survival and development. It has been seen that the ideal time to start this CPP is within the first 30 minutes of life of the newborn in any birth route, so it has been recommended that it be started in the recovery room or even in the operating room during birth by caesarean section in order to make a mark in the programming of the future physiology and behavior of the dyad.

The positive short- and long-term psychosocial, economic, environmental, and physical health effects on both maternal and infant health of adequate breastfeeding are well recognized in the literature, and yet their impact on maternal health It is not fully valued in Mexico, which maintains a very low prevalence of exclusive breastfeeding at six months of life of newborns. According to UNICEF, the prevalence of exclusive breastfeeding in Mexico is only 28.8% when in other Latin American countries it reaches 66.4%, 58.3% and 53.2%, as is the case in Peru, Bolivia and Guatemala, respectively. In 2018, Mexico is reported as having one of the lowest breastfeeding rates in the world despite having had an increase from 14.4% to 28.6% at the national level in the rate of exclusive breastfeeding.

It is very important to assess the regional conditions of our population. The cause of this low tendency to breastfeed exclusively and for a long time may have different origins in our country, such as poor or inadequate information from mothers prior to birth, false beliefs or taboos, lack of adequate support for mothers after of birth and high rates of cesarean delivery. However, it is also described that during cesarean birth it is possible to carry out actions that favor the mother-child bond and the first food to the mother's womb within the first hour of life favoring better breastfeeding. This is achieved by favoring the skin-to-skin contact between mother and baby.

However, the difficulties in ensuring that mother and baby meet in SSC may vary depending on whether it is carried out in the operating room during surgery or after it in the recovery room. It is about a procedure in which the mother-baby dyad participates as the center of care, but also all the professional support staff such as nurses, anesthesiologists and staff responsible for the care of the newborn, in addition to the obstetric staff who performs the surgery.

The foregoing leads us to ask ourselves the following research questions: Can we in our public hospitals in Mexico carry out the CPP procedure between mother and baby during cesarean births? And if so, will there be a difference in breastfeeding by Mexican women, performing skin-to-skin contact immediately even in the operating room between mother and baby in cesarean births versus if it is carried out after the surgical procedure?

ELIGIBILITY:
Inclusion Criteria: Women between 18 and 40 years of age with a single pregnancy greater than 37 weeks of gestation with an indication for cesarean section and who agree to participate in the study.

Exclusion Criteria: Patients who are minors, multiple pregnancies, or who do not agree to participate in the study.

Elimination criteria: Participants who decide not to continue with the study, who do not answer the evaluation surveys on breastfeeding or who do not return for follow-up.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding | Six months
  Feeding to the exclusive mother's breast at least six months after birth

IPD SHARING:
Plan to Share IPD: Yes
Requests for information can be requested with the principal investigator via email
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Permanently
Access Criteria: request via email

REFERENCES:
- [Background] Chien LY, Tai CJ. Effect of delivery method and timing of breastfeeding initiation on breastfeeding outcomes in Taiwan. Birth. 2007 Jun;34(2):123-30. doi: 10.1111/j.1523-536X.2007.00158.x. PMID 17542816
- [Background] Patel A, Bucher S, Pusdekar Y, Esamai F, Krebs NF, Goudar SS, Chomba E, Garces A, Pasha O, Saleem S, Kodkany BS, Liechty EA, Kodkany B, Derman RJ, Carlo WA, Hambidge K, Goldenberg RL, Althabe F, Berrueta M, Moore JL, McClure EM, Koso-Thomas M, Hibberd PL. Rates and determinants of early initiation of breastfeeding and exclusive breast feeding at 42 days postnatal in six low and middle-income countries: A prospective cohort study. Reprod Health. 2015;12 Suppl 2(Suppl 2):S10. doi: 10.1186/1742-4755-12-S2-S10. Epub 2015 Jun 8. PMID 26063291
- [Background] Stevens J, Schmied V, Burns E, Dahlen H. Immediate or early skin-to-skin contact after a Caesarean section: a review of the literature. Matern Child Nutr. 2014 Oct;10(4):456-73. doi: 10.1111/mcn.12128. Epub 2014 Apr 10. PMID 24720501
- [Background] Tully KP, Ball HL. Maternal accounts of their breast-feeding intent and early challenges after caesarean childbirth. Midwifery. 2014 Jun;30(6):712-9. doi: 10.1016/j.midw.2013.10.014. Epub 2013 Oct 26. PMID 24252711
- [Background] Lau Y, Htun TP, Lim PI, Ho-Lim S, Klainin-Yobas P. Maternal, Infant Characteristics, Breastfeeding Techniques, and Initiation: Structural Equation Modeling Approaches. PLoS One. 2015 Nov 13;10(11):e0142861. doi: 10.1371/journal.pone.0142861. eCollection 2015. PMID 26566028
- [Background] Hobbs AJ, Mannion CA, McDonald SW, Brockway M, Tough SC. The impact of caesarean section on breastfeeding initiation, duration and difficulties in the first four months postpartum. BMC Pregnancy Childbirth. 2016 Apr 26;16:90. doi: 10.1186/s12884-016-0876-1. PMID 27118118
- [Background] Sharma A. Efficacy of early skin-to-skin contact on the rate of exclusive breastfeeding in term neonates: a randomized controlled trial. Afr Health Sci. 2016 Sep;16(3):790-797. doi: 10.4314/ahs.v16i3.20. PMID 27917213
- [Background] Brimdyr K, Cadwell K, Stevens J, Takahashi Y. An implementation algorithm to improve skin-to-skin practice in the first hour after birth. Matern Child Nutr. 2018 Apr;14(2):e12571. doi: 10.1111/mcn.12571. Epub 2017 Dec 12. PMID 29230957
- [Background] Schneider LW, Crenshaw JT, Gilder RE. Influence of Immediate Skin-to-Skin Contact During Cesarean Surgery on Rate of Transfer of Newborns to NICU for Observation. Nurs Womens Health. 2017 Feb-Mar;21(1):28-33. doi: 10.1016/j.nwh.2016.12.008. PMID 28187837
- [Background] Debes AK, Kohli A, Walker N, Edmond K, Mullany LC. Time to initiation of breastfeeding and neonatal mortality and morbidity: a systematic review. BMC Public Health. 2013;13 Suppl 3(Suppl 3):S19. doi: 10.1186/1471-2458-13-S3-S19. Epub 2013 Sep 17. PMID 24564770
- [Background] Cantrill RM, Creedy DK, Cooke M, Dykes F. Effective suckling in relation to naked maternal-infant body contact in the first hour of life: an observation study. BMC Pregnancy Childbirth. 2014 Jan 14;14:20. doi: 10.1186/1471-2393-14-20. PMID 24423381
- [Background] Conde-Agudelo A, Diaz-Rossello JL. Kangaroo mother care to reduce morbidity and mortality in low birthweight infants. Cochrane Database Syst Rev. 2016 Aug 23;2016(8):CD002771. doi: 10.1002/14651858.CD002771.pub4. PMID 27552521
- [Background] Ip S, Chung M, Raman G, Chew P, Magula N, DeVine D, Trikalinos T, Lau J. Breastfeeding and maternal and infant health outcomes in developed countries. Evid Rep Technol Assess (Full Rep). 2007 Apr;(153):1-186. PMID 17764214
- [Background] Yi DY, Kim SY. Human Breast Milk Composition and Function in Human Health: From Nutritional Components to Microbiome and MicroRNAs. Nutrients. 2021 Sep 2;13(9):3094. doi: 10.3390/nu13093094. PMID 34578971
- [Background] Hauck YL, Fenwick J, Dhaliwal SS, Butt J. A Western Australian survey of breastfeeding initiation, prevalence and early cessation patterns. Matern Child Health J. 2011 Feb;15(2):260-8. doi: 10.1007/s10995-009-0554-2. PMID 20077131
- See also: Guía para la aplicación: proteger, promover y apoyar la lactancia materna en los establecimientos que prestan servicios de maternidad y neonatología - Revisión de la Iniciativa Hospitales Amigos del Niño 2018 — https://apps.who.int/iris/handle/10665/326162
- See also: Contacto Piel a Piel en cesáreasa — https://www.aeped.es/comite-nutricion-y-lactancia-materna/lactancia-materna/documentos/contacto-piel-con-piel-en-las-cesareas
- See also: Pinzamiento temprano vs tardío del cordón umbilical y contacto piel a piel inmediato en nacimientos por cesárea. — https://doi.org/10.24245/gom.v89i6.5445